CLINICAL TRIAL: NCT04675684
Title: Recovery-by-eHealth: A Complex Intervention Aiding Recovery in Patients With Depression Discharged From a Psychiatric Outpatient Clinic - a 12 Months Randomized Controlled Clinical Trial
Brief Title: Recovery-by-eHealth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Research Unit Of General Practice, Copenhagen (Other); Frederiksberg University Hospital (Other); Psychiatric Center Ballerup (Other)
Responsible Party: Principal Investigator, Anne Sofie Aggestrup, MSc, PhD student, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-20076894
Record Dates: First submitted 2020-12-03; First posted 2020-12-19 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Depression
Keywords: Recovery; Depression; Prevention; Physical health; Mental health; Randomized Controlled Trial; Mixed methods; Intersectoral collaboration
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be 1:1 randomized into either a recovery group (experimental) or a control group (no intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery-group (Experimental): The recovery group consists of:
  1. Physical, mental and social health education, advice and feedback from a health investigator.
  2. Daily self-monitoring about their mood and health in an app, Monsenso.
  3. Intersectoral collaboration between 1) Mental Health Centre Copenhagen Rigshospitalet, IAOC 2) Centre for Research and Education in General Practice, University of Copenhagen 2) Centre for Social Medicine at Frederiksberg Hospital, 3) Competence Centre for Rehabilitation and Recovery, Mental Health Centre Ballerup, and 5) Private Practicing Psychiatrists.
  Interventions: Behavioral: Recovery-group
- Control-group (No Intervention): The control group consists of usual treatment at their General Practitioner and / or Private Practicing Psychiatrist.

INTERVENTIONS:
Behavioral: Recovery-group — The complex intervention are instructions in ruminations-therapy and mindfulness, advice in healthy diets, physical - and social activities and sleep hygiene, and support in smoking cessation, alcohol counseling and medication adherence.
  Other Names: Intervention-group
  Arms: Recovery-group

SUMMARY:
This study investigates whether a complex intervention can aid recovery and prevent relapse in depression and readmissions in patients who have previously been treated for depression at a psychiatric outpatient clinic.

DETAILED DESCRIPTION:
Background: During the last seven years, our research group has collected considerable experience with conducting and contributing studies aiming to prevent relapse of depression and readmissions using a complex intervention with electronic self-monitoring in combination with feedback from health investigators. In our first study ("SAFE-I: Electronic self-monitoring with clinical feedback in depression, a feasibility study"), we used a self-monitoring system to investigate the connection between sleep and depression after discharge from a psychiatric inpatient ward to the Intensive Affective Outpatient Clinic (IAOC) in combination with weekly feedback from investigators by telephone. Patients evaluated the electronic system with a high usability score, and there was a high data entry rate. Patients gradually delayed their sleep after discharge from the psychiatric inpatient ward, and this delay of sleep was found to be related to a worsening of depression. Subsequently, we designed a Randomized Controlled Trial (RCT) ("SAFE II: Can electronic self-monitoring with closed loop feedback focusing on regulation of the sleep-wake cycle reduce relapse of depression after discharge from a psychiatric ward") that included patients before discharge from a psychiatric inpatient ward and in the early faces of their stay at IAOC, and followed them for four weeks. Patients were randomized to one group using electronic self-monitoring with feedback from health investigators focusing on self-reported data, and another group that in addition to the electronic self-monitoring was guided to attain signals to the circadian clock to stabilize the, sleep-wake cycle (diet, daylight exposure, sleep, and behavioral motivation towards social function and physical activity). In all, 103 patients were included in the trial (last patient visit 22-12-2020). From the qualitative data in this study, we found that patients expressed a feeling of support and safety by participating in the study. They especially felt that the electronic self-monitoring with continuous feedback from investigators provided them with an important reflection on their activity and mental health. The depression severity decreased significantly in both groups, comparable to what was found in the SAFE-I study. Readmission rates were low in both groups (7.8 %). However, the study lacked an independent evaluation of the implementation of the health interventions, i.e. process evaluation. Users were not involved in the study's design. The SAFE-studies found that feedback from investigators is deemed critical for a positive outcome, a finding supported by reviews of studies using electronic self-monitoring in combination with feedback from investigators for patients with depression. This proposed trial comprise further development based on experiences from these studies.

Objective: Recovery-by-eHealth investigates whether a complex intervention can aid recovery and prevent relapse in depression and readmissions in patients who have previously been treated for depression at a psychiatric outpatient clinic.

Design: A randomized controlled trial. Participants will be 1:1 randomized into either an recovery-group or a control-group.

Intervention: Participants allocated to the recovery-group will make daily self-monitoring about their physical, mental and social health in an app for one week in total each month. At the end of these weekly periods a health investigator will phone the patients to provide feedback. Additional calls are allowed when needed. Patients allocated to the control-group will follow their usual treatment at their general practitioner and/or private practice psychiatrist.

The project will be an intersectoral collaboration between 1) Mental Health Centre Copenhagen Rigshospitalet, Intensive Affective Outpatient Clinic 2) Centre for Research and Education in General Practice, University of Copenhagen 2) Centre for Social Medicine at Frederiksberg Hospital, 3) Competence Centre for Rehabilitation and Recovery, Mental Health Centre Ballerup, and 5) Private Practicing Psychiatrists.

Inclusion criteria:

* Age > 18 years
* Treated for depression at the IAOC for minimum 6 months and with a planned continued treatment in primary health care

Exclusion criteria:

* Psychotic depression at inclusion
* Dementia or other organic brain disorders
* Alcohol substance abuse that is expected to interfere with the study procedures
* INSPIRE-O score > 65 at inclusion

Primary outcome:

• Personal recovery self-assessed by the Brief INSPIRE-O scale

Secondary outcomes:

* Number of relapses of depression blindly assessed by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
* Depressive symptoms self-assessed by the Hamilton Depression Rating 6-item Scale (Ham-D6)
* Well-being self-assessed by the WHO-5 scale
* Recovery support self-assessed by the INSPIRE scale

Explorative outcomes:

* Adherence to medication according to Medicine Adherence Rating Scale (MARS)
* Rate of hospital re-admissions
* Perceived stress according to Cohen's Perceived Stress Scale (PSS)
* The Perseverative Thinking Questionnaire (PTQ) to assess repetitive negative thinking and anxiety
* Rate of biochemistry: C-Reactive Protein (CRP; mg/dL), total-cholesterol (mg/dL), Low-Density Lipoprotein cholesterol (LDL; mg/dL), Low-Density Lipoprotein cholesterol (HDL; mg/dL), triglyceride (mg/dL), thyrotropin (TSH; mIU/L), vitamin-D (nmol/L) and HbA1c, oxidative stress, and hair cortisol
* Rate of Body Mass Index (BMI)
* Rate of blood pressure
* Rate of psychiatric readmissions in a five-year follow-up period after ending the study
* Rate of connection to the labor market in a five-year follow-up period after ending the study

Qualitative data will be used to support the quantitative outcomes.

Trial size: 130 participants.

Time schedule: The trial has been submitted for regulatory approvals November 2020, the first participant will be included August 2021, the expected last follow-up of the last participant will be August 2024. Data will be analyzed and published from August 2023 till August 2024, and we expect to submit the first manuscript December 2023.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Treated for depression at the IAOC for minimum 6 months and with a planned continued treatment in primary health care

Exclusion Criteria:

* Psychotic depression at inclusion
* Dementia or other organic brain disorders
* Alcohol substance abuse that is expected to interfere with the study procedures
* INSPIRE-O score > 65 at inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Personal recovery self-assessed by the Brief INSPIRE-O scale | 12 months
  Difference between the two groups in return to personal recovery from baseline until 12 months after baseline measured whit Brief INSPIRE-O's 5-item self-rated measure of personal recovery.

SECONDARY OUTCOMES:
Recovery support self-assessed by the INSPIRE scale | 12 months
  Difference between the two groups in return to recovery support from a clinician/worker from baseline until 12 months after baseline measured with Brief INSPIRE's 5-item self-rated measure of recovery support from a clinician/worker.
Depressive symptoms self-assessed by the Hamilton Depression Rating 6-item Scale (Ham-D6) | 12 months
  Difference between the two groups in return to symptoms of depression from baseline until 12 months after baseline measured with Hamilton Depression Rating Scale consisting of 6 items. Total scores from zero (no depression) to 22 (most severe depression).
Wellbeing self-assessed by the WHO-5 scale | 12 months
  Difference between the two groups in return to wellbeing from baseline until 12 months after baseline measured with WHO-5's wellbeing self-assessed scale consisting of 5 items.
Number of relapses of depression blindly-assessed by the Mini International Neuropsychiatric Interview | 12 months
  Difference between the two groups in return to number of relapses of depression from baseline until 12 months after baseline measured with a short, structured clinical diagnostic interview based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).

OTHER OUTCOMES:
Adherence to medication according to Medicine Adherence Rating Scale (MARS) | 12 months
  Difference between the two groups in return to medication adherence from baseline until 12 months after baseline from patients interviews and patient records (explorative outcome).
Rate of hospital re-admissions | 12 months
  Difference between the two groups in return to rate of hospital re-admissions during the project period from patient interviews and patient records (explorative outcome).
Perceived stress self-assessed by the Perceived Stress Scale (PSS) | 12 months
  Difference between the two groups in return to perceived stress according to Cohen's Perceived Stress Scale (PSS) from baseline and until 12 months after baseline (explorative outcome).
Repetitive negative thinking and anxiety self-assessed by the Perseverative Thinking Questionnaire (PTQ) | 12 months
  Difference between the two groups in return to repetitive negative thinking and anxiety according to the Perseverative Thinking Questionnaire (PTQ) from baseline and until 12 months after baseline (explorative outcome).
Blood level | 12 months
  Difference between the two groups in return to the following blood levels: C-Reactive Protein (CRP), total-cholesterol, Low-Density Lipoprotein (LDL), Low-Density Lipoprotein (HDL), and triglyceride (mg/dL) from baseline until 12 months after baseline from patient records (explorative outcome).
Weight (kg) | 12 months
  Difference between the two groups in return to weight (kg) from baseline until 12 months after baseline. The participants weight (kg) and height (meter) will be combined to calculate their Body Mass Index (kg/m^2) (explorative outcome).
Height (meter) | 12 months
  Difference between the two groups in return to height (meter) from baseline until 12 months after baseline. The participants weight (kg) and height (meter) will be combined to calculate their Body Mass Index (kg/m^2) (explorative outcome).
Blood pressure | 12 months
  Difference between the two groups in return to blood pressure (mm Hg) from baseline until 12 months after baseline (explorative outcome).
Blood level | 12 months
  Difference between the two groups in return to Thyrotropin (TSH; mIU/L) from baseline until 12 months after baseline (explorative outcome).
Blood level | 12 months
  Difference between the two groups in return to Vitamin D (nmol/L) from baseline until 12 months after baseline (explorative outcome).
Blood level | 12 months
  Difference between the two groups in return to Hemoglobin A1c (HbA1c; mmol/mol) from baseline until 12 months after baseline (explorative outcome).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.psykiatri-regionh.dk/nid-group